CLINICAL TRIAL: NCT06723925
Title: Neonatal Screening of Biotinidase Deficiency: Genotype-phenotype Correlation and Clinical Follow-up of Patients Identified At the Regional Centre for Neonatal Screening of Endocrine-Metabolic Diseases in Bologna
Brief Title: Neonatal Screening of Biotinidase Deficiency: Genotype-phenotype Correlation and Clinical Follow-up
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: BiotiPed
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Biotinidase Deficiency
Keywords: Biotinidase Deficiency
MeSH Terms: conditions — Biotinidase Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Retro-prospective, single-centre, observational study conducted at the Endocrine-Metabolic Diseases Center of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy.

The study involves children born in Emilia-Romagna region, Italy, from January 2016 to December 2020 with biotinidase deficiency identified through Neontal Screening at the Endocrine-Metabolic Diseases Center of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy. The primary aim of this study is to assess the incidence of biotinidase decificiency in this cohort of patients and the possible correlation between the genotype and the biochemical and clinical phenotype of this cohort of patients.

DETAILED DESCRIPTION:
The study consists of the retrospective collection and analysis of clinical, biochemical and genetic data of pediatric patients who were taken in charge for Biotinidase Deficiency at the Endocrine-Metabolic Diseases Center of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy, following Neonatal Screening positivity.

For this cohort of patients, a clinical evaluation is planned annually after the diagnosis of Biotinidase Deficiency for the identification of possible long-term complications. A clinical follow-up of at least 36 months is expected.

According to clinical practice, parents of pediatric patients with Biotinidase Deficiency identified through Neonatal Screening will undergo molecular genetic analysis for specific familial mutations of the BTD gene, but will not be followed up.

ELIGIBILITY:
INCLUSION CRITERIA:

FOR PEDIATRIC PATIENTS

* Neonatal Screening test result of Residual biotinidase Enzyme Activity <50% carried out from January 2016 to December 2019 at the Endocrine-Metabolic Diseases Center of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy;
* Neonatal Screening test result of Residual biotinidase Enzyme Activity <30% carried out from January 2020 to December 2020 at the Endocrine-Metabolic Diseases Center of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy;
* Obtaining informed consent from parents or legal guardian of pediatric patients.

FOR PARENTS

* Being a parent of a paediatric patient enrolled in the study;
* Availability of parental data;
* Obtaining informed consent.

EXCLUSION CRITERIA:

* Subjects with known chromosomal abnormalities or complex syndromes.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with Biotinidase Deficiency (and their parents) identified through Neonatal Screening from January 2016 to December 2020 at the Endocrine-Metabolic Diseases Center of the Pediatrics Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
BTD gene mutation | baseline
  allele1, allele2 mutations
Residual biotinidase Enzymatic Activity | baseline
  percentage %
Biotin replacement therapy | baseline
  mg/die
Presence of Sintomatology | annually after the diagnosis of Biotinidase Deficiency up to 3 yaers
  ocular, dermatological, neuropsychiatric symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Rita Ortolano, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy